CLINICAL TRIAL: NCT05760339
Title: Preoperative Intermittent Fasting Versus Carbohydrate Loading to Reduce Insulin Resistance: a Randomised Controlled Trial
Brief Title: Intermittent Fasting Versus Carbohydrate Drinks Before Surgery
Acronym: PRINCESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: European Society of Anaesthesiology and Intensive Care (Other)
Responsible Party: Principal Investigator, B Preckel, Prof. dr., Amsterdam UMC, location AMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRINCESS trial
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Perioperative Care; Intermittent Fasting; Carbohydrate Loading; Preoperative Fasting; Orthopedic Surgery; Insulin Resistance
Keywords: Perioperative Care; Carbohydrate Loading; Orthopedic Surgery; Insulin Resistance; HOMA-IR; Time Restricted Feeding
MeSH Terms: conditions — Intermittent Fasting; Insulin Resistance | interventions — Diet, Carbohydrate Loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Time-restricted feeding (Experimental): Subjects will follow a daily time-restricted feeding regimen consisting of an 8h ad libitum eating period and a 16h water fasting period during the last two weeks before surgery, followed by routine preoperative fasting before surgery.
  Interventions: Behavioral: Time-restricted feeding
- Carbohydrate loading (Active Comparator): Subjects will follow their usual diet in the pre-surgical weeks and will receive a maltodextrin beverage on the evening before surgery, as well as two hours before induction of anaesthesia
  Interventions: Dietary Supplement: Carbohydrate loading
- Control group (No Intervention): Subjects will continue their usual diet and proceed with standard preoperative fasting (i.e., eat up until 6 hours and take clear liquids up until 2 hours before induction of anaesthesia).

INTERVENTIONS:
Behavioral: Time-restricted feeding — Subjects in the will be instructed to follow a TRF regimen consisting of a daily 8h ad libitum eating period and 16h water fasting period during the last 2 weeks before surgery. Participants will be encouraged to begin their eating period at 08:00h and end it at 16:00h, since the metabolic benefits of TRF appear to be considerably more pronounced when the eating period starts early in the day.
  Arms: Time-restricted feeding
Dietary Supplement: Carbohydrate loading — Subjects will continue their usual diet and will receive two quantities of a clear beverage containing 12.5 g/100 mL maltodextrin (50 kCal/100 mL, pH 5.0); 800 mL at 22.00h on the evening before surgery and 400 mL two hours before anaesthesia induction.
  Arms: Carbohydrate loading

SUMMARY:
The purpose of this study is to investigate whether time-restricted feeding, a form of intermittent fasting, before surgery improves insulin resistance around the time of surgery, compared to carbohydrate drinks and standard fasting before surgery.

DETAILED DESCRIPTION:
Patients in the Time-Restricted Feeding (TRF) group will follow a daily TRF regimen consisting of an 8h ad libitum eating period and a 16h water fasting period during the last two weeks before surgery, followed by routine preoperative fasting before surgery.

Patients in the CarboHydrate Loading (CHL) group will follow their usual diet in the pre-surgical weeks and will receive a maltodextrin beverage on the evening before surgery, as well as two hours before induction of anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective orthopaedic surgery;
* Intermediate, major or complex surgery according to the Surgical Outcome Risk Tool (SORT; http://www.sortsurgery.com/) severity of surgery classification;
* Scheduled for surgery at least 17 days from the date of screening;
* Motivated to follow a time restricted feeding regimen.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* History of diabetes mellitus;
* History of feeding or eating disorders;
* History of delayed gastric emptying or gastro-oesophageal reflux
* Active malignancy
* Patients classified as ASA IV by the attending anaesthetist;
* BMI < 18.5 or ≥ 35;
* Outpatient or day case surgery;
* Palliative surgery;
* Participation in another clinical trial that is interfering with the procedures or outcomes of the PRINCESS trial;
* Patients unable to fully comply to study needs (e.g. legally incapable patients or patients unable to communicate in Dutch).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance on postoperative day 1 | Postoperative day 1
  Insulin resistance according to the updated homeostasis model assessment of insulin resistance (HOMA2-IR)

SECONDARY OUTCOMES:
Difference in HOMA2-IR | From baseline to day of surgery, from baseline to postoperative day 1 and from day of surgery to postoperative day 1.
  This is a calculated value between two timepoints, in contrary to the primary outcome that solely measures postoperative insulin resistance. The preoperative HOMA2-IR and the postoperative HOMA2-IR are used to determine whether there has been a change (increase or decrease) of the insulin resistance.
Beta-cell function | The day of surgery and the first postoperative day
  The beta-cell function is based on the updated HOMA2 model. In addition to glucose and insulin, C-peptide measurements will be done to calculate HOMA2-B.
Patient wellbeing | During the two weeks preoperatively, until one day postoperatively
  Patient wellbeing during and after the intervention and on the first postoperative day is measured by combining the five-level EuroQol five-dimensional questionnaire (EQ-5D-5L) utility score (change in scores 1-5 over 5 domains, 1 is best and 5 is worst), and the Quality of Recovery-15 (QoR-15) score (0-150, 0 is the worst and 150 is the best recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Hermanides, MSc, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request following the completion of the trial and publication of the final manuscript. The shared data may include de-identified data that contains individual-level data collected during the trial. Researchers seeking data access must submit a research proposal and analysis plan outlining objectives, methodology, and relevance. If applicable, approval by a medical ethics research committee is required. Proposals will be reviewed to ensure that the request aligns with scientific and ethical standards, and data access will be granted under a data use/sharing agreement that stipulates the terms and conditions for data usage.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After completion of the trial and publication of the final manuscript.
Access Criteria: Researchers seeking data access must submit a research proposal and analysis plan outlining objectives, methodology, and relevance. If applicable, approval by a medical ethics research committee is required. Proposals will be reviewed to ensure that the request aligns with scientific and ethical standards, and data access will be granted under a data use/sharing agreement that stipulates the terms and conditions for data usage.

REFERENCES:
- [Derived] Stobbe AY, de Klerk ES, van Wilpe R, Kievit AJ, Choi KF, Preckel B, Hollmann MW, Hermanides J, van Stijn MFM, Hulst AH. Study protocol of the PRINCESS trial-PReoperative INtermittent fasting versus CarbohydratE loading to reduce inSulin resiStance versus standard of care in orthopaedic patients: a randomised controlled trial. BMJ Open. 2025 Jan 21;15(1):e087260. doi: 10.1136/bmjopen-2024-087260. PMID 39842917